CLINICAL TRIAL: NCT00984750
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Effect of 6-month Acetylcarnitine Therapy on Arterial Blood Pressure, Lipid and Metabolic Profile, and Kidney Function in Hypertensive Patients With Type 2 Diabetes on Background Simvastatin Therapy
Brief Title: Acetyl-L-Carnitine in Type 2 Diabetes
Acronym: DIABASI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Leadiant Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIABASI; 2007-005925-31 (EudraCT Number)
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Acetylcarnitine; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Statin and acetyl-L-carnitine
  Interventions: Drug: acetyl-L-carnitine/statin (simvastatin)
- 2 (Placebo Comparator): Statin and placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: acetyl-L-carnitine/statin (simvastatin) — acetyl-L-carnitine: 4 tablets of 500 mg a day
  simvastatin: 10 to 20 mg/day as deemed clinically appropriate and according to tolerability
  Arms: 1
Drug: placebo — placebo: 4 tablets of 500 mg a day simvastatin: 10 to 20 mg/day as deemed clinically appropriate and according to tolerability
  Arms: 2

SUMMARY:
Decreased insulin sensitivity (or insulin resistance) is a major risk factor for type 2 diabetes mellitus and renal and cardiovascular disease. It is the key component and, possibly, a pathogenetic factor of the metabolic syndrome - a clustering of arterial hypertension, obesity, impaired glucose tolerance, dyslipidemia, coagulation abnormalities, albuminuria and increased cardiovascular risk - that may precede or accompany type 2 diabetes.

Insulin function and the abnormalities associated with insulin resistance, may have a major role in preventing type 2 diabetes and, in the long-term, diabetes micro- and macrovascular complications. Carnitine is involved in lipids and carbohydrates metabolism and acetyl-L-carnitine (ALC), an intramitochondrial carrier of acylic group, may modulate cell fuel substrate utilization. Studies found that carnitine may improve insulin sensitivity and glucose disposal in healthy subjects and in patients with type 2 diabetes. A recent study found that a primed constant infusion of acetyl-L-carnitine (ALC) may increase glucose utilization in type 2 diabetic patients, possibly restoring the glycogen synthase activity.

In a previous pilot study in healthy subjects with decreased insulin sensitivity, the investigators found that 6-month treatment with Acetyl-L-Carnitine - an ester of l-carnitine - improved the glucose disposal rate, taken as a marker of insulin sensitivity. Amelioration of insulin sensitivity was associated with a significant and clinically relevant reduction in systolic blood pressure without appreciable changes in diastolic blood pressure. Whether blood pressure reduction reflected the amelioration of insulin sensitivity or, rather, a direct, specific effect of Acetyl-L-Carnitine is still unknown.The antihypertensive effect ensued progressively and slowly waned after treatment withdrawal as documented by a slow and progressive increase in blood pressure levels toward baseline levels over the recovery period. This finding provided convincing evidence that blood pressure reduction throughout the observation period was not explained by a "trial effect", but reflected a true treatment effect. Blood pressure was a secondary efficacy variable of the study and mechanisms underlying the antihypertensive effect of Acetyl-L-Carnitine (such as reduced peripheral resistances, decreased cardiac output, increased artery compliance and/or enhanced sodium excretion), in this population were not assessed.

Acetyl-L-Carnitine was well tolerated in all of the patients and may provide a novel therapeutic tool for the treatment of arterial hypertension, and of dyslipidemia and could be safely used in people with type 2 diabetes.

Thus, the investigators designed a prospective, randomized, double-blind, placebo-controlled trial to investigate whether Acetyl-L-Carnitine added-on stable and standardized blood pressure and lipid lowering therapy may help further improving control of hypertension and dyslipidemia and, therefore, decreasing the overall cardiovascular risk in hypertensive patients with type 2 diabetes.

DETAILED DESCRIPTION:
BACKGROUND Arterial hypertension, in particular systolic hypertension, is a common component of the metabolic syndrome, a syndrome of hypertension, abdominal obesity, dyslipidemia, impaired glucose tolerance and increased urinary albumin excretion sustained by decreased tissue sensitivity to insulin (insulin resistance). It affects 80 to 90% of people with type 2 diabetes and is the strongest risk factor for macrovascular and microvascular complications of diabetes, such as myocardial infarction, stroke, peripheral artery disease, nephropathy and retinopathy. Despite multi-drug therapy, reduction of systolic blood pressure to normal range is seldom achievable in people with type 2 diabetes. Moreover, due to increased vascular stiffness, reducing systolic blood pressure may decrease diastolic blood pressure to the extent that diastolic myocardial perfusion is impaired and the risk of ischemic event increased. Thus, availability of drugs that may help controlling systolic hypertension without appreciably affecting diastolic blood pressure would have major clinical implications.

In addition to arterial hypertension, dyslipidemia is also a component of the metabolic syndrome that is almost invariably observed in people with type 2 diabetes and remarkably contributes to the excess cardiovascular risk in this population. HMGCoA inhibition by statin therapy, significantly ameliorates hypercholesterolemia, but only marginally affects the concomitant hypertriglyceridemia (probably the most typical feature of increased insulin resistance) and fails to significantly reduce the circulating levels of serum lipoprotein(a), one of the strongest predictors of coronary and cerebrovascular events in type 2 diabetics. Thus, availability of drugs that may help achieving a more effective amelioration of dyslipidemia in this population might also have important clinical implications .

In an ongoing study in healthy subjects with decreased insulin sensitivity, we found that 6-month treatment with acetylcarnitine - an ester of l-carnitine - improved the glucose disposal rate, taken as a marker of insulin sensitivity. Amelioration of insulin sensitivity was associated with a significant and clinically relevant reduction in systolic blood pressure without appreciable changes in diastolic blood pressure. Whether blood pressure reduction reflected the amelioration of insulin sensitivity or, rather, a direct, specific effect of acetylcarnitine is still unknown.

Previous studies also found that L-carnitine added on background simvastatin therapy, marginally affected serum cholesterol, but remarkably reduced serum triglyceride and lipoprotein (a) levels. Whether amelioration of insulin resistance may explain at least in part this effect is unclear.

Finally, all available clinical studies consistently showed that acetyl carnitine is a well tolerated drug that can be safely used in humans. Experimental evidence is also available that l-carnitine may improve statin-associated myotoxicity.

AIMS Primary To asses the effect of 6-month therapy with acetylcarnitine compared to placebo on systolic blood pressure in 228 patients with type 2 diabetes, arterial hypertension and dyslipidemia on stable background antihypertensive, hypoglycemic, and lipid lowering therapy.

Secondary

A.To asses the effect of treatment on:

* diastolic and pulse pressure
* serum triglycerides and apolipoprotein(a)
* HOMA index (calculated during data analyses), serum insulin, leptin, adiponectin (pending on the findings on the other efficacy variables)
* blood glucose, serum cholesterol (total, HDL and LDL), non-esterified fatty acids (NEFA), lipoproteins A and and uric acid
* 2-hours post oral load blood glucose profile
* high density C-reactive protein (hsCRP)
* urinary albumin excretion and estimated creatinine clearance (calculated during data analyses)
* cardiac output, peripheral resistances or large artery compliance (as assessed by echocardiography in a representative subgroup)
* 24 hour sodium excretion and sodium fractional clearance, in a representative subgroup
* need for concomitant therapy with antihypertensive, hypoglycemic, and lipid lowering agents

B.To assess whether the observed changes in systolic, diastolic or pulse pressures and in lipid or metabolic profile correlate with the concomitant changes in markers of insulin sensitivity.

C.To monitor systolic/diastolic blood pressure and other clinical/laboratory parameters evaluated during the study two months after Acetyl-L-Carnitine therapy or Placebo withdrawal in patients completing the study and maintained on the same background medications.

DESIGN The study will be a prospective, randomized, double-blind, placebo-controlled, multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >40 years old;
* High-risk subjects with type 2 diabetes (WHO criteria);
* High blood pressure (systolic blood pressure >140 mmHg or with concomitant antihypertensive treatment stable since at least 3 months);
* Serum creatinine concentration <1.5 mg/dl;
* Patients legally able to give written informed consent to the trial (signed and dated by the patient);
* Written informed consent.

Exclusion criteria:

* Uncontrolled diabetes (glycated hemoglobin >11%);
* Acute cardiovascular events over the last 3 months;
* Specific contraindications or history of hypersensitivity to the study drugs;
* Previous history of allergy or intolerance, or evidence of immunologically-mediated renal disease, systemic diseases, cancer;
* Drug or alcohol abuse;
* Any chronic clinical conditions that may affect completion of the trial or confound data interpretation;
* Pregnancy or lactating;
* Women of childbearing potential without following a scientifically accepted form of contraception;
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial;
* Evidence of an uncooperative attitude;
* Any evidence that patient will not be able to complete the trial follow-up.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Arterial blood pressure and dyslipidemia | Basal, 15th day, 30th day, 3rd and 6th month

CONTACTS AND LOCATIONS:
Overall Officials: Piero Ruggenenti, MD, Study Director — Mario Negri Institute for Pharmacological Research
Locations (5):
- Italy (5):
  - Hospital "Azienda Ospedaliera Ospedali Riunitidi Bergamo" Unit of Diabetology, Bergamo, Bergamo
  - Hospital "Azienda Ospedaliera di Treviglio e Caravaggio" Ambulatory of Diabetology, Ponte San Pietro, Bergamo
  - Clinical Research Center for Rare Diseases "Aldo and Cele Daccò", Ranica, Bergamo
  - Hospital "Azienda Ospedaliera di Treviglio-Caravaggio"Unit of Diabetology and Metabolic Diseases, Romano di Lombardia, Bergamo
  - Hospital "Azienda Ospedaliera di Treviglio-Caravaggio" Unit of Diabetology and Metabolic Disease, Treviglio, Bergamo